CLINICAL TRIAL: NCT04653519
Title: Accuracy and Reproducibility of Virtually Guided Minimally Invasive Tooth Preparations Using Reverse Engineering (Controlled Clinical Trial)
Brief Title: Accuracy and Reproducibility of Virtually Guided Minimally Invasive Tooth Preparations Using Reverse Engineering
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, yara attia, Assistant Lecturer of Fixed Prosthodontics, Fayoum University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0155-09/2020
Record Dates: First submitted 2020-11-19; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Marginal Adaptation of Fixed Dental Prosthesis
Keywords: Minimally invasive tooth preparations; Reverse engineering; Virtually guided tooth preparation; Digital assessment of tooth preparation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtually guided minimally invasive preparation (Experimental)
  Interventions: Device: Virtually guided minimally invasive preparation

INTERVENTIONS:
Device: Virtually guided minimally invasive preparation — Intraoral virtually guided minimally invasive design with an occlusal reduction of 1.5mm, axial reduction will be performed with 6 degrees axial taper and a circumferential chamfer margin of 0.5mm in width and 0.5mm coronal to the gingival margin. A milled guiding occlusal resin template of the teeth will be checked for fitting then fixed using spot etching and will be used to guide the amount of axial reductions and taper degree.

SUMMARY:
The aim of the study is to assess and reproduce standardized virtually guided minimally invasive tooth preparations using digitally designed occlusal template, compared to its reference virtual preparation using a computer aided 3-dimensional (3-D) analysis, and to investigate the effect of these preparations on absolute marginal discrepancy of 3 unit monolithic translucent zirconia FPD using a computer aided 3-D analysis.

DETAILED DESCRIPTION:
Ten patients with missing mandibular first molar will receive a three-unit full contour monolithic zirconia FPD. Each patient case will receive two modes of preparation as in the previous in-vitro study: virtually guided tooth preparation using occlusal resin template to assist the intraoral preparation and the reference virtual tooth preparation. Each participant's preparation will be evaluated using diagnostic dental software and will be compared to a reference digital virtual preparation using 3-D mesh processing reverse engineering metrology software.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a missing lower first mandibular molar.
* Good oral hygiene with no signs of periapical pathology or periodontal disease (periodontal screening index 0-1) and with compliance to perform strict oral hygiene measures.
* Well-aligned abutment teeth with similar mesio-distal (M-D) and bucco-lingual (B- L) dimensions; (2nd premolar: M-D 7.8 mm ±1, B-L 8.7 mm ±1), (2nd molar: M-D 10.73±1, B-L 10.5 mm ±1).
* Abutment teeth with an adequate occluso-gingival height where (2nd premolar: 8.4 mm ±1, 2nd molar 7mm ±1), and adequate edentulous span length (9.5 mm±1); for an appropriate connector area of at least 9 mm.
* Absence of parafunctional habits (clinching, bruxism).

Exclusion Criteria:

* Bad oral hygiene.
* Advanced periodontitis, gingivitis, or recession.
* Abutments with subgingival restorations, root caries.
* Parafunctional habits.
* Undergoing orthodontic treatment.
* Obvious dentition malalignment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the virtually guided tooth preparation accuracy | 1 month
  Each scan data of virtually guided preparations will be uploaded to a 3D mesh processing reverse engineering software, then superimposed against the reference virtual preparation using the software's best fit matching algorithm tool. Superimposed 3D data files will be sectioned into 5 different 2D planes: buccolingual, mesiodistal, transverse occlusal, transverse middle, and transverse gingival. Differences will be assessed both qualitatively and quantitively to measure deviations. Quantitative assessment will be expressed with a sign: (+) indicating external deviation or (-) indicating internal deviation. The deviation (+ or -) will be numerically described with mean and standard deviation. Qualitative assessment will be through a color-coded mapping of superimposed images where discrepancies between each test specimen and reference file will be expressed with yellow range of color lines indicating external deviations and cyan range of color lines indicating internal deviations
3-D Evaluation of absolute marginal discrepancy using reverse engineering | 1 month
  Four scans will be performed using a calibrated laboratory scanner: each 3D printed master cast with 2 preparations designs, external & intaglio surfaces of monolithic zirconia 3-unit FPDs, monolithic zirconia 3-unit FPDs after it has been seated on each preparation design. The 3D point clouds of all 4 scans will be obtained in STL format. The 3D data of the FPD retainers will be registered to the data obtained from the external surface of the crown using registration module in reverse engineering software. The 3D data of the virtual seating of the intaglio & external surfaces on the preparations will be obtained & margins of the FPD retainers & preparations will be extracted. The software's construct cross-sectional cloud circular command to divide the preparation evenly into curves. Every curve will intersect with the outer edge of the ceramic retainer & margin design of the preparation at 2 points. Distance between these 2 points will be recorded (absolute marginal discrepancy)

CONTACTS AND LOCATIONS:
Overall Officials: Yara H Attia, M.Sc, Principal Investigator — Faculty of Dentistry, Fayoum University, Egypt; Samir I Bakry, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Sanaa H Abd El Kader, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt